CLINICAL TRIAL: NCT06304519
Title: Identifying the Optimal Patient-Specific Dynamic Ankle-Foot Orthosis Bending Stiffness in an Evidence-Based Manner That Can be Implemented by Clinical Providers
Brief Title: Identifying the Optimal Dynamic Ankle-Foot Orthosis Bending Stiffness for Individuals Post-Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 1986626-1
Record Dates: First submitted 2024-02-23; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: ankle-foot orthosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dynamic ankle-foot orthosis — customized, carbon fiber, passive ankle-foot orthosis

SUMMARY:
Ankle braces are commonly prescribed to individuals who have suffered a stroke to help their ankle joints work properly, which allows these individuals to walk better. Currently, there are no standardized guidelines to follow when choosing which brace is best for an individual. Prior work has shown that customizing the level of assistance that these braces provide based on each individual's level of ankle impairment improves the individuals' walking function more than their current brace. The next important step is to fine-tune the customization and work to develop a set of guidelines that can be used by clinicians to help them prescribe the right brace for each patient's needs. The purpose of this study is to test different levels of assistance provided by the brace to determine the optimal customization method. Additionally, this study aims to begin to create a guide to help clinicians choose the best brace for each individuals' needs. To accomplish this goal, individuals will walk with a brace under five different assistance level conditions. The individual's walking function, performance on clinical measures, and response to questionnaires will be examined to determine both the optimal brace for each individual and hopefully identify clinical tools that can be used to guide prescription of the brace. This study is a major step towards developing effective, standardized prescription guidelines that optimize walking of individuals post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (> 6 months post-stroke)
* been prescribed an AFO by a clinician
* have plantar flexor strength deficits (unable to complete at least 25 standing heel-raises
* have at least 5 degrees of passive dorsiflexion range of motion (as measured during the clinical evaluation in Visit 1).

Exclusion Criteria:

* Those that will not be included in this study are individuals with 1) Evidence of cerebellar stroke on clinical MRI, 2) Other neurologic conditions in addition to stroke, 3) Sensorimotor neglect, 4) Inability to walk outside the home prior to the stroke, 5) Total joint replacement or orthopedic problems in the lower limbs or spine that limit walking, 6) Coronary artery bypass graft or myocardial infarction within past 3 months, 7) Unexplained dizziness in last 6 months, 8) Inability to communicate with investigators, 9) Lack of decisional capacity.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Mechanical Cost of Transport of the Lower Extremities | Day 2
Sagittal plane ankle moment during stance | Day 2
Sagittal plane ankle angle during stance | Day 2
Self-selected walking speed | Day 2
a candidate set of clinical outcome measures | Day 2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware STAR Campus, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No